CLINICAL TRIAL: NCT05503355
Title: A Phase I/II Dose Escalation and Expansion Study of BST-236 Plus Venetoclax in Patients With Newly Diagnosed Acute Myeloid Leukemia Unfit for Intensive Induction Chemotherapy
Brief Title: A Phase I/II Dose Escalation and Expansion Study of BST-236 Plus Venetoclax in Patients With Unfit Newly Diagnosed AML
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: BioSight Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BST005
Record Dates: First submitted 2022-08-14; First posted 2022-08-16 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2022-08

CONDITIONS: AML, Adult
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): BSR-236 + venetoclax
  Interventions: Drug: BST-236; Drug: venetoclax

INTERVENTIONS:
Drug: BST-236 — In part 1: During the induction (in combination with venetoclax), the BST-236 doses are:
  In cohort 1 - 2.3 g/m2/d X6 days In cohort 2 - 2.3 g/m2/d X6 days In cohort 3 - 4.5 g/m2/d X6 days In cohort 4 - 4.5 g/m2/d X6 days In cohort 5 - 4.5 g/m2/d X6 days In part 1: During maintenances (for responding patients) the BST-236 dose- 4.5 g/m2/d X6 days In part 2, the dose chosen as safe and efficacious for induction in part 1 will be used
Drug: venetoclax — In part 1: During the induction (in combination with BST-236), the venetoclax doses are:
  In cohort 1 - 200 mg QD X 7 days In cohort 2 - 400 mg QD X 7 days In cohort 3 - 200 mg QD X 7 days In cohort 4 - 400 mg QD X 7 days In cohort 5 - 200 mg QD X 14 days In part 2, the dose chosen as safe and efficacious for induction in part 1 will be used
  Other Names: Venclevta

SUMMARY:
An open label multi centre study to assess the safety and efficacy of BST-236 in combination with venetoclax in adult patients unfit for standard therapy with newly diagnosed Acute Myeloid Leukemia (AML) Part 1 of the study will define the maximal tolerate dose of the combination treatment, while part 2 will expend the chosen dose, to assesses efficacy and safety of this combination.

All patients will receive 2 induction courses with both BST-236 and venetoclax, responding patients will then be followed with up to 3 maintenance courses with BST-236 alone. Patients will be followed for 1 year in the study and additional 1 year in post study follow-up

ELIGIBILITY:
Inclusion Criteria:

1. Adult ≥18 years of age
2. Diagnosis of AML (de-novo AML or AML secondary to MDS or secondary to exposure to potentially leukemogenic therapies or agents)
3. Not eligible for standard induction chemotherapy
4. Peripheral white blood cell (WBC) count of <25,000/μL
5. Creatinine clearance ≥45 mL/min
6. AST and/or aALT ≤2.5 X ULN)
7. Total bilirubin ≤1.5 x ULN
8. ECOG PS of:

   * 0 to 2 for patients ≥75 years of age
   * 0 to 3 for patients <75 years of age
9. Women of reproductive potential must have a negative serum pregnancy test within 48 hours of Study Day 1

Exclusion Criteria:

1. Patient has acute promyelocytic leukemia
2. Any previous treatment for AML
3. Patient has a known history of myeloproliferative neoplasm (MPN)
4. Patient has known active central nervous system (CNS) involvement with AML
5. Use of an investigational drug within 5 half-lives (or 30 days in case the half-life is unknown) prior to Study Day 1
6. Previous BM/stem cell transplantation (SCT)
7. Previous treatment for MDS with cytarabine, hypomethylating agents, or venetoclax
8. For Part 1 only - use of known strong or moderate CYP3A inducers within 7 days prior to Study Day 1
9. Patient has consumed grapefruit, grapefruit products, Seville oranges (including marmalade containing Seville oranges), or starfruit within 3 days prior to Study Day 1
10. Patient has a malabsorption syndrome or other condition that precludes enteral route of drug administration
11. Uncontrolled systemic fungal, bacterial, or viral infection (defined as ongoing signs/symptoms related to the infection without improvement despite appropriate antibiotics or other treatment)
12. Any medical or surgical condition, presence of clinical safety laboratory abnormalities, or psychiatric illness that may preclude safe and complete study participation based on the Investigator's judgment.
13. Diagnosis of malignant disease other than AML within the previous 12 months
14. Diagnosis of myeloid sarcoma as a sole manifestation of AML
15. Unstable angina, significant cardiac arrhythmia, or New York Heart Association (NYHA) Class IV CHF
16. History of allergic reactions attributed to compounds of similar chemical composition as BST-236 and/or cytarabine and/or venetoclax.
17. Surgical procedure, excluding central venous catheter placement or other minor procedures (e.g. skin biopsy) in the 14 days prior to enrollment

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-08-17 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicity and maximal tolerated dose for part 2 | Up to day 42
In part 2: | Up to day 42 of second induction
  Complete remission rate

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Northwestern Memorial Hospital, Chicago, Illinois
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - University of Virginia Cancer Center, Charlottesville, Virginia